CLINICAL TRIAL: NCT06248541
Title: The Effect of Low-Level Laser Therapy in Carpal Tunnel Syndrome: A Randomized, Single-Blinded, Placebo-Controlled Trial
Brief Title: The Effect of Low-Level Laser Therapy in Carpal Tunnel Syndrome
Acronym: KaLi-CTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK-NR:35-255 ex 22/23
Record Dates: First submitted 2024-01-25; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: CTS
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Therapeutics; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: treatment with low-level laser therapy (Experimental): Patient gets treated with a low-level laser (wavelength of 620 - 640nm) two times a day for 3 weeks.
  Interventions: Device: treatment with low-level laser therapy
- Group 2: treatment with conventional light diodes (Placebo Comparator): Patient gets treated with conventional light diodes two times a day for 3 weeks.
  Interventions: Device: treatment with conventional light diodes

INTERVENTIONS:
Device: treatment with low-level laser therapy — low-level laser therapy (wavelength of 620 - 640nm)
  Arms: Group 1: treatment with low-level laser therapy
Device: treatment with conventional light diodes — conventional light diodes
  Arms: Group 2: treatment with conventional light diodes

SUMMARY:
Carpal tunnel syndrome (CTS) is a chronic compression of the median nerve, which can lead to symptoms such as nocturnal pain and paresthesia in the area innervated by the median nerve. The affected patients also describe discomfort and hypoesthesia in the nerve supply area. Due to the COVID (Coronavirus disease) pandemic, CTS operations have been postponed and delayed. A promising and safe alternative for improving CTS-related symptoms appears to be non-invasive, non-thermal low-level-laser therapy. As a possible conservative, alternative method, low-level-laser therapy has the potential to enable patients with CTS to improve their disease-related symptoms or at least to alleviate the symptoms until the indicated CTS operation (carpal tunnel release).

The aim of this randomized, single-blind, placebo-controlled clinical trial is to investigate the influence of 3 weeks of low-level-laser therapy on the symptoms typical of CTS in patients with surgery-indicated carpal tunnel syndrome and its influence on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Existing written consent of the participating person after informed consent.
* The patient is capable of giving consent.
* Isolated surgery-induced CTS
* CTS patients with pain (NRS between 2 and 6) and/or paresthesia and/or nocturnal pain that has been present for at least 3 months (pain reported using the "Numerical Rating Scale for Pain" (NRS) between 0 and 10).
* Compliance with 3 weeks of cold light therapy.

Exclusion Criteria:

* Absence of informed consent
* Patients under 18 years or over 80 years
* Patients from protected groups as well as people who are not able to personally give consent
* Participation in other clinical trials within the last 4 weeks before the start of the study
* traumatic and atraumatic median nerve lesions/damage/narrowing
* Previous operations in the area innervated by the median nerve or in the area of the affected upper extremity/hand
* CTS recurrence of the affected hand
* Thenar atrophy of the affected hand
* Nerve diseases that affect the upper extremity including the hand (e.g. polyneuropathy)
* Cervical radiculopathy C6/C
* Osteoarthritis of the affected hand (e.g. rhizarthrosis)
* Arthritis of the affected hand
* Metabolic diseases that have an influence on the sensory or function of the hand
* Vascular diseases affecting the upper extremity or hand (e.g. Raynaud's syndrome)
* other compressions or injuries of the median nerve (e.g. thoracic outlet syndrome, scalene syndrome, pronator teres syndrome)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain: at rest (Numerical Rating Scale for Pain, NRS) | baseline, after 3 weeks, after 6 weeks
  Pain at rest (NRS), scale 0-10, higher score indicates worse pain
Pain:movement pain (Numerical Rating Scale for Pain, NRS) | baseline, after 3 weeks, after 6 weeks
  Pain at activity (NRS), scale 0-10, higher score indicates worse pain
Pain: Night pain (Numerical Rating Scale for Pain, NRS) | baseline, after 3 weeks, after 6 weeks
  Pain over night (NRS), scale 0-10, higher score indicates worse pain
Health-related quality of ife (SF-36 ) | baseline, after 3 weeks, after 6 weeks
  Health-related quality of life assessed by SF-36 questionnaire, scores 0-100 for each SF-36 subdomains (out of eight subdomains), higher scores indicates better qualitiy of life
Hand function (Quick-DASH) | baseline, after 3 weeks, after 6 weeks
  Hand function assessed by Quick-DASH (Disabilities of Arm, Shoulder and Hand) questionnaire, 19-95, lower scores indicates better hand function
Hand function and CTS severity (Boston CTS Syndrome Questionnaire) | baseline, after 3 weeks, after 6 weeks
  Hand function and CTS severity assessed by Boston CTS Syndrome Questionnaire (BCTQ)), score range 19 - 95, a higher score indicates lower hand function and more severe CTS symptoms

SECONDARY OUTCOMES:
Demographic patient data: smoking status | 1 day (baseline)
  smoking status
Demographic patient data: previous illnesses | 1 day (baseline)
  History of Previous illnesses
Medication (painkillers / immunosuppressives) | baseline, after 3 weeks, after 6 weeks
  Medication taken by patients during the study (painkillers: yes/no, immunosuppressives: yes/no)
Hofmann-Tinel sign (positive / not positive) | baseline, after 3 weeks, after 6 weeks
  Hofmann-Tinel sign (positive / not positive)
Phalen test (positive / not positive) | baseline, after 3 weeks, after 6 weeks
  Phalen test (positive / not positive)
2-point discrimination | baseline, after 3 weeks, after 6 weeks
  2-point discrimination test, distance in millimeters
Sensitivity (Semmes-Weinstein monofilament) | baseline, after 3 weeks, after 6 weeks
  Sensitivity (Semmes-Weinstein monofilament)
Hand strength / grip strength" | baseline, after 3 weeks, after 6 weeks
  measured with Jamar dynamometer
Nerve conduction velocity of the median nerve | baseline
  Nerve conduction velocity of the median nerve (extracted from hospital intern database if available)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Hecker, MSc. Dr., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria